CLINICAL TRIAL: NCT02420769
Title: Color Doppler of CL and Uterine Artery With Serum Progesterone and CA125 in Threatened Abortion
Brief Title: Corpus Luteum and Uterine Artery Doppler With Serum P and CA125 in Threatened Abortion
Acronym: CLCA125
Status: Completed | Type: Observational
Sponsor: Nesreen Abdel Fattah Abdullah Shehata (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Sponsor-Investigator, Nesreen Abdel Fattah Abdullah Shehata, Assisstant professor of Obstetrics and Gynecology, Beni-Suef University
Organization: Beni-Suef University (Other)
Other Study IDs: Beni-Suef 9
Record Dates: First submitted 2015-04-05; First posted 2015-04-20 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Threatened Abortion
Keywords: CA 125; Progesterone; Doppler; Corpus Luteum
MeSH Terms: conditions — Abortion, Threatened

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Threatened abortion: Pregnant patients > 8 weeks gestation coming to the ANC clinic with mild vaginal bleeding but healthy viable intrauterine pregnancy. Vaginal color doppler for uterine artery and corpus luteum together with serum progesterone and CA125 will be assessed.

SUMMARY:
The purpose of this study is to determine whether assessing color doppler of corpus luteum and uterine artery is useful in predicting patients who will complete pregnancy. The investigators will add to this the usefulness of serum progesterone and CA125 in prediction.

DETAILED DESCRIPTION:
The introduction of Doppler ultrasound in obstetrics has allowed evaluating hemodynamic characteristics from the first trimester of pregnancy. For example, Kurjak et al.,in one of the first studies using transvaginal pulsed-wave Doppler ultrasound in early pregnancies, identified the uterine arteries in 100% of the patients. The flow blood of the corpus luteum was identified in 75% patients. The measures obtained by Doppler ultrasonography that may have prognostic value to the evolution of pregnancy include uteroplacental blood flow, also known as trophoblastic flow. Jaffe et al. reported that abnormal Doppler findings were associated with a significantly higher prevalence of complicated pregnancies, among women with abnormal Doppler findings, 43% ended in miscarriage, whereas among women with normal findings only 1.4% of women miscarried.Progesterone plays a crucial role in the maintenance of pregnancy. In the presence of sufficient progesterone levels during pregnancy, lymphocytes synthesize a mediator called progesterone induced blocking factor (PIBF), which is anti-abortive in mice . Besides inducing secretary changes in the endometrium and supporting early pregnancy, it modulates the maternal immune response to prevent fetal rejection and relaxes the uterine smooth muscles .CA-125, well-known as a tumor marker for epithelial ovarian cancer , is a high molecular weight glycoprotein that is produced not only by ovarian cancer, but also by nonovarian tumors, normal epithelia of the peritoneum, the endometrium, the fallopian tube, and the ovary. Because CA-125 is also produced by the endometrium, some authors suggest that CA-125 can be used as a marker for endometrial receptivity in patients undergoing IVF . Its role as a predictor for pregnancy outcome is controversial .

ELIGIBILITY:
Inclusion Criteria:

* patients with pregnancy between 8 to 20 weeks of gestation,
* who were diagnosed with threatened abortion.

Exclusion Criteria:

* patients with multiple pregnancies,
* molar pregnancy,
* ectopic pregnancy,
* amenorrhea with different etiologies of pregnancy,
* maternal history of systemic diseases and uterine anatomic abnormalities
* patients who did not have their outcome data through week 20 of gestation due to relocation.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant females >8 weeks but < 20 weeks gestation. They are presenting with a complaint of threatened abortion to our outpatient ANC clinic.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Viable fetus (According to WHO viable fetus >500 gm or > 20 weeks) | from 20 weeks till 21 weeks gestation
  The investigators will assess how many patients in both groups reached viability of fetus. According to WHO viable fetus >500 gm or > 20 weeks.

SECONDARY OUTCOMES:
Resistance index of uterine artery and corpus luteum | from 8 weeks till 20 weeks
  Vaginal color doppler of uterine artery and corpus luteum for all pregnant patients in the study at first visit in ANC clinic .
serum CA125 and progesterone | from 8 weeks till 20 weeks gestation
  serum CA125 and progesterone will be done for all pregnant patients at first visit in ANC clinic

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen A Shehata, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kurjak A, Crvenkovic G, Salihagic A, Zalud I, Miljan M. The assessment of normal early pregnancy by transvaginal color Doppler ultrasonography. J Clin Ultrasound. 1993 Jan;21(1):3-8. doi: 10.1002/jcu.1870210103. PMID 8478442
- [Background] Jaffe R, Dorgan A, Abramowicz JS. Color Doppler imaging of the uteroplacental circulation in the first trimester: value in predicting pregnancy failure or complication. AJR Am J Roentgenol. 1995 May;164(5):1255-8. doi: 10.2214/ajr.164.5.7717242.
- [Background] Kalinka J, Szekeres-Bartho J. The impact of dydrogesterone supplementation on hormonal profile and progesterone-induced blocking factor concentrations in women with threatened abortion. Am J Reprod Immunol. 2005 Apr;53(4):166-71. doi: 10.1111/j.1600-0897.2005.00261.x. PMID 15760377
- [Background] Potdar N, Konje JC. The endocrinological basis of recurrent miscarriages. Curr Opin Obstet Gynecol. 2005 Aug;17(4):424-8. doi: 10.1097/01.gco.0000175363.20094.bd. PMID 15976551
- [Background] Miranda S, Litwin S, Barrientos G, Szereday L, Chuluyan E, Bartho JS, Arck PC, Blois SM. Dendritic cells therapy confers a protective microenvironment in murine pregnancy. Scand J Immunol. 2006 Nov;64(5):493-9. doi: 10.1111/j.1365-3083.2006.01841.x. PMID 17032241
- [Background] Bast RC Jr, Feeney M, Lazarus H, Nadler LM, Colvin RB, Knapp RC. Reactivity of a monoclonal antibody with human ovarian carcinoma. J Clin Invest. 1981 Nov;68(5):1331-7. doi: 10.1172/jci110380. PMID 7028788
- [Background] Phocas I, Sarandakou A, Rizos D, Dimitriadou F, Mantzavinos T, Zourlas PA. Tumour-associated antigens, CEA, CA 125 and SCC in serum and follicular fluid of stimulated and unstimulated cycles. Eur J Obstet Gynecol Reprod Biol. 1994 Apr;54(2):131-6. doi: 10.1016/0028-2243(94)90252-6. PMID 8070597
- [Background] Miller KA, Deaton JL, Pittaway DE. Evaluation of serum CA 125 concentrations as predictors of pregnancy with human in vitro fertilization. Fertil Steril. 1996 Jun;65(6):1184-9. doi: 10.1016/s0015-0282(16)58336-8. PMID 8641495
- [Background] Chryssikopoulos A, Mantzavinos T, Kanakas N, Karagouni E, Dotsika E, Zourlas PA. Correlation of serum and follicular fluid concentrations of placental protein 14 and CA-125 in in vitro fertilization-embryo transfer patients. Fertil Steril. 1996 Oct;66(4):599-603. doi: 10.1016/s0015-0282(16)58574-4. PMID 8816623
- [Result] Gustavo Romero-Gutiérrez, Antonio Abraham Huebe-Martínez, Immer Amaral-Navarro, Armando Saú Ruiz-Treviño. Doppler Ultrasound Assessment in Women with Threatened Abortion, Clinical Medicine Research. Vol. 2, No. 3, 2013, pp.24-28. doi: 10.11648/j.cmr.20130203.11
- [Derived] Shehata NAA, Ali HAA, Hassan AEGMA, Katta MA, Ali ASF. Doppler and biochemical assessment for the prediction of early pregnancy outcome in patients experiencing threatened spontaneous abortion. Int J Gynaecol Obstet. 2018 Nov;143(2):150-155. doi: 10.1002/ijgo.12631. Epub 2018 Aug 31. PMID 30058068